CLINICAL TRIAL: NCT05703620
Title: REducing Sympathetic Activity Through Ultrasound-based Renal deneRvation in Excessive Cardiovascular Risk populaTions - the RESURRECT Trial. A Pilot Proof-of-concept and Safety Study With the Paradise Denervation System
Brief Title: REducing Sympathetic Activity Through Ultrasound-based Renal deneRvation in Excessive Cardiovascular Risk populaTions.
Acronym: RESURRECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Perth Hospital (Other)
Collaborators: ReCor Medical, Inc. (Industry)
Responsible Party: Principal Investigator, Professor Markus Schlaich, Principal Investigator, Royal Perth Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHC20190025
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Chronic Kidney Diseases; Heart Failure; End Stage Renal Disease
Keywords: Renal Denervation; Sympathetic Nervous System
MeSH Terms: conditions — Renal Insufficiency, Chronic; Heart Failure; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chronic Kidney Disease (Experimental): Renal Denervation
  Interventions: Device: Renal Denervation
- Heart Failure (Experimental): Renal Denervation
  Interventions: Device: Renal Denervation
- End stage renal disease (Experimental): Renal Denervation
  Interventions: Device: Renal Denervation

INTERVENTIONS:
Device: Renal Denervation — All eligible participants receive ultrasound based renal denervation to both kidneys on all eligible vessels

SUMMARY:
The is a non-randomized pilot trial, open-label evaluation of the physiologic response of native kidney denervation using the Paradise denervation system in CKD, End Stage Renal Disease (ESRD), and Heart failure (HF)

DETAILED DESCRIPTION:
There is unequivocal evidence for an important contribution of increased renal sympathetic nerve activity to cardiovascular (CV) morbidity and mortality in high risk patient cohorts with CKD, ESRD and HF. The availability of a highly effective catheter-based ultrasound device to selectively target renal nerves provides a potential unique opportunity to improve CV outcomes in these patients, a proposition that now needs to be tested in initial pilot trials and subsequent appropriately designed randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria:

* Both Male and female patients
* Ages between 18-75 years of age
* Individual is competent and willing to provide written, informed consent to participate in this clinical study with either

  * CKD stage 3a/b or
  * ESRD on stable renal replacement therapy or
  * Mild to moderate heart failure with reduced ejection fraction

Exclusion Criteria:

* Ineligible anatomy
* Prior treatment with other devices for hypertension including but not limited to ROX Coupler (ROX Medical) , Mobius stent, and/or the CVRx (CVRx Inc) barostimulator device.
* Individual has experienced a myocardial infarction, unstable angina, or a cerebrovascular accident within 3 months of the screening visit.
* Documented history of chronic active inflammatory bowel disorders such as Crohn's disease or ulcerative colitis.
* Individual has clinically significant cardiac structural valvular disease, unless corrected by a properly functional prosthetic valve
* Individual has been admitted for inpatient hospitalization for decompensated HF in the previous month
* Female participants of childbearing potential must have a negative pregnancy test prior to treatment.
* Individual has a known, unresolved history of drug use or alcohol dependency, lacks the ability to comprehend or follow instructions, or would be unlikely or unable to comply with study follow-up requirements.
* Individual is currently enrolled in another investigational drug or device trial. Note: For the purpose of this protocol, participants involved in extended follow-up trials for products that were investigational but are currently commercially available are not considered enrolled in an investigational trial.
* Individual has a disease or condition (aside from CKD, ESRD, and HFrEF) that may limit their life expectancy to < 1 year.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-10-08 (Actual); Primary Completion 2025-05-18 (Estimated); Study Completion 2026-05-18 (Estimated)

PRIMARY OUTCOMES:
Reduction in renal sympathetic nerve activity | BASELINE TO 3 MONTHS
  Spillover results
Reduction in renal sympathetic nerve activity | BASELINE TO 12 MONTHS
  Muscle Sympathetic Nerve Activity (MSNA)

SECONDARY OUTCOMES:
Blood Pressure | Baseline to 36 months
  Changes in systolic and diastolic blood pressures

CONTACTS AND LOCATIONS:
Overall Officials: Markus Schlaich, Principal Investigator — Royal Perth Hospital
Locations (1):
- Royal Perth Hospital, Perth, Western Australia, Australia